CLINICAL TRIAL: NCT00979381
Title: Study to the Humoral and Cellular Immunoresponse After Influenza Vaccination in Patients With Metastasized RCC or GIST Treated With a Tyrosine Kinase Inhibitor(Sunitinib or Sorafenib)
Brief Title: Study of the Immunoresponse in Patients Treated With a Tyrosine Kinase Inhibitor
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: C.M.L. van Herpen, UMCN St Radboud
Other Study IDs: UMCNONCO20084
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2009-09

CONDITIONS: Renal Cell Carcinoma; GIST
Keywords: sunitinib; sorafenib; immune response
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Patients with metastasized renal cell carcinoma or GIST who have been treated with sunitinib or sorafenib for at least 4 weeks
  Interventions: Biological: influenza vaccine
- 2: patients with metastasized RCC who did not receive a systemic treatment for their RCC (nephrectomy is allowed)
  Interventions: Biological: influenza vaccine
- 3: healthy volunteers
  Interventions: Biological: influenza vaccine

INTERVENTIONS:
Biological: influenza vaccine — influenza vaccination

SUMMARY:
In this study the researchers investigate the influence of the tyrosine kinase inhibitors sunitinib and sorafenib, on the normal humoral and cellular immuno response to influenza vaccination in patients with metastases of renal cell carcinoma or a GIST.

DETAILED DESCRIPTION:
When cure is not longer possible, cancer patients enter the palliative phase. For many types of cancer several treatment options are available. The goal of this treatment is to prolong survival, but maintenance or even improvement of quality of life is of equal importance. The currently available systemic treatment options consist of conventional cytotoxic therapy, hormonal therapy, immunotherapy and the so-called targeted therapies. Combinations of these therapies are also being used. Targeted therapy concerns the application of a new class of drugs that are specifically directed against one or more well-defined molecular targets that are relevant for carcinogenesis, cell cycle regulation, tumour progression, metastasis, tumour angiogenesis and/or apoptosis. Today, the most successful drugs in this class are directed against the vascular endothelial growth factor (VEGF) and the epidermal growth factor receptor (EGFR). There is an explosive development ongoing in this field and many new drugs become available that have new targets or inhibit a combinations of targets. Meanwhile, targeted therapy has shown efficacy in many types of cancer and is registered for several indications. The toxicity profile of targeted therapies is still largely unknown, and the aetiology of many known side effects has not been clarified. At the moment, three targeted therapies that are directed against VEGF are registered and used in the Netherlands: Sunitinib (Sutent®) and Sorafenib (Nexavar ®) both oral drugs and Bevacizumab (Avastin®), an intravenously drug. Clinical experience and some mouse studies show that targeted therapies could have a negative effect on the immune response. This can be of great influence on patients who are treated with this type of drug.

Especially because these drug will be used chronically and sometimes for years and infections can have a large influence on the health and quality of life of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastasized renal cell carcinoma or GIST who have been treated with sunitinib or sorafenib for at least 4 weeks, or patients with metastasized RCC who did not receive a systemic treatment for their RCC (nephrectomy is allowed)
* Patients who are indicated for influenza vaccination and and have been summoned for this vaccination by their GP
* age ≥18 years (for the healthy volunteers: age≥ 60 years)
* signed Informed Consent Form

Exclusion Criteria:

* patients with an identified immunodeficiency disorder
* patients that have been treated with corticosteroids in the past 2 weeks or who are still using these (except for a short period <10 days)
* patients that are treated with immunotherapy in the last year (ex. interferon-alpha of IL-2) or who have received another form of targeted therapy (ex. bevacizumab).
* patients with symptoms of influenza at the time of vaccination
* patient with an allergy for chicken-eggwhite

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with metastasized renal cell carcinoma or GIST who have been treated with sunitinib or sorafenib for at least 4 weeks, or patients with metastasized RCC who did not receive a systemic treatment for their RCC (nephrectomy is allowed)
  * Patients who are indicated for influenza vaccination and and have been summoned for this vaccination by their GP
  * healthy volunteers who have been summoned by theire GP to receive a influenza vaccin
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2008-10; Primary Completion 2008-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
cellular and humoral immune response | 1 year

SECONDARY OUTCOMES:
times the influenza virus occurs | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: C.M.L. van Herpen, MD, Phd, Principal Investigator — UMCN st Radboud
Locations (1):
- University Medical Center Nijmegen st Radboud, Nijmegen, Netherlands